CLINICAL TRIAL: NCT04818138
Title: Canadian Atopic Dermatitis Cohort for Translational Immunology and Imaging (CACTI) With a Nested BROadband vs Narrowband photoTherapy for Eczema (BRONTE) Randomized Controlled Trial
Brief Title: BROadband vs Narrowband photoTherapy for Eczema Trial Nested in the CACTI Cohort
Acronym: BRONTE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of funding period.
Sponsor: Women's College Hospital (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); University of British Columbia (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Aaron Drucker, Scientist, Women's College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CACTI
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Atopic Dermatitis; Skin Diseases; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Skin Diseases; Eczema

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Narrowband UVB (Active Comparator): Narrowband UVB phototherapy (full body) administered three times weekly according to individual clinical protocols.
  Interventions: Device: Narrowband UVB phototherapy
- Broadband UVB (Active Comparator): Broadband UVB phototherapy (full body) administered three times weekly according to individual clinical protocols.
  Interventions: Device: Broadband UVB phototherapy

INTERVENTIONS:
Device: Narrowband UVB phototherapy — Narrowband UVB phototherapy (full body) administered three times weekly according to individual clinical protocols.
  Other Names: NBUVB
  Arms: Narrowband UVB
Device: Broadband UVB phototherapy — Broadband UVB phototherapy (full body) administered three times weekly according to individual clinical protocols.
  Other Names: BBUVB
  Arms: Broadband UVB

SUMMARY:
Atopic dermatitis (eczema) is a complicated skin condition. In fact, it represents many different underlying problems. These include abnormalities in the skin barrier, the immune system and the ability to handle different bacteria. Despite many recent gains in the understanding of eczema, a lot needs to be learned. There is little evidence to select between some of the older treatments that are available now. Even the newest targeted therapy does not clear most patients' skin. In order to improve the understanding of eczema, how to treat it now, and to enable discovery of new treatments, the investigators plan to enroll patients into a large study at three centres in Canada (University of Toronto, McGill University and University of British Columbia). The study is called the Canadian Atopic Dermatitis Cohort for Translational Immunology and Imaging (CACTI). In this study, the investigators will collect data on how severe participants' eczema is and what treatments they use. For participants who give permission, the investigators will collect blood and skin biopsy samples to study the mechanisms underlying their disease. The investigators will test to see which form of phototherapy (Broadband or Narrowband Ultraviolet B phototherapy) works best for eczema in a randomized clinical trial. The investigators will also use advanced imaging techniques to visualize the skin.

This trial registry entry, including the description of the treatment arms and outcomes, refer to the nested BROadband vs Narrowband photoTherapy for Eczema clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Atopic dermatitis according to the Hanifin and Rajka criteria.
2. Validated Investigator Global Assessment score of 3 or 4 out of 4
3. Eczema Area and Severity Index (EASI) score ≥7.1
4. Moderate to severe disease as above despite an adequate trial of topical therapy.

Exclusion Criteria:

1. Treatment with phototherapy or oral systemic immune-modulating agents (cyclosporine, methotrexate, azathioprine, mycophenolate) less than 30 days before baseline.
2. Treatment with systemic biologic (dupilumab) or experimental therapeutic less than 90 days before baseline.
3. Current treatment with oral or intramuscular corticosteroids within 30 days prior to baseline. Topical, intralesional or inhaled corticosteroids are allowed.
4. Participating in a clinical trial assessing an investigational agent for atopic dermatitis (topical, systemic or device) within 90 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Mean change in the Eczema Area and Severity Index (EASI) from baseline | Week 12
  The EASI measures clinical signs of atopic dermatitis. The minimum value is 0, the maximum is 72. Higher scores indicate worse disease.

SECONDARY OUTCOMES:
Proportion of patients achieving a validated Investigator Global Assessment (vIGA) score of 0 or 1 with a ≥ 2 point improvement from baseline | Week 12
  The IGA measures clinical signs of atopic dermatitis. The minimum value is 0, the maximum is 4. Higher scores indicate worse disease.
Mean change in the Patient Oriented Eczema Measure (POEM) from baseline | Week 12
  The POEM measures symptoms of atopic dermatitis. The minimum value is 0, the maximum is 28. Higher scores indicate more frequent symptoms.
Mean change in the Peak Pruritus Numeric Rating Scale (PP-NRS) from baseline | Week 12
  The PP-NRS measures itch. The minimum value is 0, the maximum is 10. Higher scores indicate worse itch.
Mean change in the Dermatology Life Quality Index (DLQI) from baseline | Week 12
  The DLQI measures skin-specific quality of life. The minimum value is 0, the maximum is 30. Higher scores indicate worse impact on quality of life.
Mean change in the Recap of atopic eczema (RECAP) | Week 12
  The RECAP measures atopic dermatitis control. The minimum value is 0, the maximum is 28. Higher scores indicate worse atopic dermatitis control.

OTHER OUTCOMES:
Mean change in EuroQol-5D-5L (EQ5D-5L) from baseline | Week 12
  The EQ5D is an instrument to assess overall health state. Values are normalized to normative populations. Lower scores indicate worse overall health.
Mean change in body surface area (BSA) from baseline | Week 12
  BSA is the percentage (0-100) of skin involved with atopic dermatitis lesions.
Change in the patient global assessment scale from baseline | Week 12
  Patient global assessment measures the patient's perception of their overall atopic dermatitis severity (clear, almost clear, mild, moderate, severe).
Withdrawal from phototherapy due to adverse events | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Aaron M Drucker, Principal Investigator — Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The full protocol for the CACTI study and nested BRONTE trial will be made publicly available.
  The anonymized participant-level dataset and statistical code for the BRONTE trial will be made available to qualified investigators upon request.